CLINICAL TRIAL: NCT06721897
Title: Effectiveness of a Prehabilitation Program on Clinical, Functional and Psychological Variables in Candidates for Hip or Knee Arthroplasty Surgery.
Brief Title: Effectiveness of a Prehabilitation Program for Hip or Knee Arthroplasty Surgery.
Acronym: Preoperative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Irene María Lopera Pareja (Other)
Collaborators: University of Jaén (Other)
Responsible Party: Sponsor-Investigator, Irene María Lopera Pareja, Principal Investigator, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 003_sep24 - PI2 - Prehabilitac
Record Dates: First submitted 2024-11-28; First posted 2024-12-06 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Prehabilitation; Knee Osteoarthritis; Hip Osteoarthritis; Physical Therapy Modalities
Keywords: prehabilitation; knee osteoarthritis; hip osteoarthritis; physiotherapy preoperative
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group (IG) will undergo a 6-week prehabilitation program for total hip/knee replacement surgery. Once the surgery is complete, they will follow the same rehabilitation program proposed for the control group.
  Interventions: Other: Prehabilitation Program
- Control Group (Experimental): The control group (CG) will carry out a post-operative physiotherapy program in addition to a home exercise program that will be shown by the physiotherapist before hospital discharge.
  Interventions: Other: Non prehabilitation Program

INTERVENTIONS:
Other: Prehabilitation Program — A prehabilitation programme supervised by a physiotherapist in a ward is proposed, with a frequency of 3 sessions/week on alternate days lasting 30-45 min/session, in addition to a daily physical exercise programme at home.
  The programme will consist of a warm-up, strength exercises with progressive loads, proprioception, balance, cardiovascular training aimed at functional work and a cool-down.
  The home programme will be complementary to the supervised programme, which will consist of daily sessions of 20-30 min of flexibility and proprioception exercises.
  The same prehabilitation protocol will be proposed for those patients awaiting total hip and knee replacement surgery.
  Arms: Intervention Group
Other: Non prehabilitation Program — The control group (CG) will carry out a post-operative physiotherapy program in addition to a home exercise program that will be shown by the physiotherapist before hospital discharge.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
We live in an increasingly aging society in which the incidence of osteoarticular diseases increases, among which osteoarthritis (OA) stands out. OA is a degenerative disorder of the different components of the joint leading to a progressive destruction of the same. The hip and knee being the most affected joints, OA presents multiple symptoms such as pain, stiffness and functional limitation, also causing psychological disorders such as anxiety, depression, quality of sleep and poor perception of quality of life. Conventional treatment is aimed at alleviating symptoms, but when conservative therapies fail in the more advanced stages of the disease, total joint replacement surgery or arthroplasty is the therapeutic option of choice. Strength physical exercise (PE) and aerobic training have been shown to be effective in OA, obtaining positive effects on the symptoms and on variables that deteriorate this disease. The concept of pre-habilitation or preoperative rehabilitation has been shown through other studies in different pathologies (cardiopulmonary and musculoskeletal) to have positive effects at a clinical and functional level, however, the planning of a pre-habilitation protocol in hip or knee arthroplasty is still controversial.

The purpose of this study is to determine the effect that a prehabilitation program will produce and its possible usefulness in those subjects who are waiting for a hip or knee arthroplasty. It is expected to find favorable results that support this therapy when it comes to reducing postoperative recovery times, functional capacity and other psychological variables of interest.

This powerful tool could represent a non-pharmacological and non-invasive therapy, as well as being useful and economical in the management of patients with OA in advanced stages.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hip OA stage I-III of the Tönnis classification or diagnosis of knee OA stage I-IV of the Ahlbäck classification
* Patients requiring hip/knee arthroplasty surgery
* Signed informed consent
* Obtaining a score equal to or greater than 8 repetitions in the Sit to Stand test
* Patients with the ability to walk without technical aids or in need of some help (up to two canes or a walker)

Exclusion Criteria:

* Cognitive deficit/Dementia states
* Cancer processes
* Associated vascular and inflammatory pathologies
* Associated neurological pathologies
* Contraindications to physical exercise

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring Quality of life | Start of the study and week 24
  SF-12 Health Questionnaire: This is a valid instrument for measuring health-related quality of life (HRQoL). The SF-12 is a reduced version of the SF-36 questionnaire, consisting of a subset of 12 items from the SF-36, selected by multiple regression, including 1 or 2 items from each of the 8 domains of the SF-36. From the information obtained from these 12 items, the SF-12 physical and mental summary measures are obtained as the only assessments. The assessments vary between 0 (no quality of life) and 100 (maximum quality of life).

SECONDARY OUTCOMES:
Lower limb functionality | Start of study, week 6, week 9 and week 24
  Time Up and Go Test: Evaluates functional capacity through walking and balance, as well as its probable disorders in an elderly subject. It consists of timing the time to perform the following test: get up from a chair and walk at a normal pace a distance of 3 meters, have the person turn around, walk back to the chair and sit down again (6 meters in total). This test has three levels of interpretation: normal/independent (if the subject takes less than 20 seconds), slight risk of falling (between 20-29 seconds) and high risk of falling or dependency (values greater than 30 seconds). If the patient requires technical aids, this must be indicated on the data sheet. Two attempts are made and the best time is chosen.
Lower limb functionality | Start of study, week 6, week 9 and week 24.
  Sit to Stand Test: This consists of counting the number of repetitions that the person gets up and sits down in a chair for 30 seconds. To do this, the subject will be seated in the chair in a posture that allows him to place his feet flat on the floor and separated at the height of his hips, with his knees bent at just over 90º. He will be told that his arms will remain crossed in front of his chest during the test. If the subject cannot lift anything in this position, he will be allowed certain adaptations (hands on his legs or on technical aids) noting said adaptations together with the number of repetitions. Each age range and sex has variable intervals of number of repetitions, although scores below 8 indicate a high risk of falls in both sexes.
Strength | Start of study, week 6, week 9 and week 24 (end of intervention).
  Manual dynamometer: A low-cost, noninvasive method for assessing muscle strength. It is performed using a portable pressure algometer "Pain Test FPN 100" (Wagner Instruments, USA). Three attempts are made, each separated by 30 seconds. The manual dynamometer is a valid and reliable tool for measuring muscle strength, with an ICC between moderate and high (0.55 and 0.85) depending on the muscle group evaluated.
Strength | Start of the study, week 6, week 9 and week 24 (end of the intervention)
  1RM - Brizky's formula: Test to assess endurance in multi-joint exercises. The most common application of this test is to assess changes in muscle strength during training periods. A simple and cost-effective test that does not require expensive equipment, hence its high use. In the case of estimating 1RM in patients with OA, it will be calculated using the indirect Brzycki method in the contralateral (unaffected) limb. To do this, the patient must perform between 6-10 repetitions of each exercise to be assessed with a fixed load that is not very high (5kg). After obtaining the number of repetitions performed with that load, the Brzycki formula will be applied (lifted weight/(1.0278-(0.0278*number of repetitions)) which will give us the value of 1 RM with the established load. In the event that the exercise to be performed cannot be done with a weight, a set of mini-bands of different resistances (expressed in kilograms) will be used with which this same test will be performed.
Level of perceived exertion | From the start of the prehabilitation program until 6 weeks (end of the prehabilitation program)
  Modified Borg scale: Adapted from the classic perceived exertion (RPE) scale, the modified Borg scale is used to measure dyspnea and the intensity of the entire exercise session. It has a gradation from 0 to 10, where 0 represents the absence of dyspnea/rest and 10 is the maximum degree of dyspnea/exertion, so that the subject can indicate the level of perceived exertion subjectively during the training session.
Intensity of Pain | Start of the intervention, week 6, week 9 and week 24.
  Numeric Pain Rating Scale- NPRS: This is a scale for assessing pain intensity in a unidimensional manner. This subjective scale consists of 11 items (0-10) where 0 corresponds to no pain and 10 to maximum pain, so that the user can communicate the level of pain he or she has or perceives while performing the task.
Psychological aspects | Start of intervention, week 6 and week 24.
  Goldberg Anxiety and Depression Scale (GADS): It is a useful tool to guide towards the diagnosis of anxiety or depression (or both) in addition to discriminating and sizing the intensities of each of them. It is composed of 2 subscales (anxiety subscale and depression subscale) with nine questions each. In the anxiety subscale (questions 1-9) a minimum of 2 questions from the first four questions must be answered affirmatively in order to continue with the subscale. In the case of the depression subscale (questions 10-18) it is sufficient to answer affirmatively one question from questions 10-13 in order to proceed to answer the rest. The total score varies from 0-18 points so that for the anxiety subscale the cut-off points are 4 points or more and 2 or more points for the depression subscale, the maximum score being 9 points for each subscale.
Sleep Quality | Start of the intervention and week 24
  Pittsburgh Scale: This is an instrument for assessing sleep quality. It is made up of 24 items (although only 19 are taken into account for obtaining data) divided into 7 dimensions. Each dimension has 4 values on a scale of 0 to 3. The total ICSP score is obtained from the sum of the 7 dimensions, which ranges from 0 to 21 points (the higher the score, the worse the sleep quality).
Analgesic consumption | Start and week 6.
  Analgesic consumption: An activity diary is used to mark the days of the week that drugs are taken for OA pain relief. Therefore, values are measured from 0-7 days/week
Therapeutic adherence | Start of the intervention and week 6.
  Therapeutic adherence: continuous quantitative metric variable. It was collected through a registration sheet provided at the beginning of the trial. It recorded the days per week of physical activity (0-7 days/week) as well as the duration of daily physical activity, taking values of number of hours/week.
Treatment expectations and therapeutic satisfaction | 24/48 hours post-surgery
  Nottingham Health Profile: Self-administered questionnaire designed to measure health perception and assess the extent to which health problems affect daily life activities. It consists of two parts, the first consisting of 38 questions that explore 6 dimensions of health (energy, pain, physical mobility, emotional state, sleep and social isolation). The second part consists of 7 questions about the functional limitations that the health problem causes in seven situations of daily life (work, housework, social life, family life, sexual life, hobbies and free time). Each question is answered with a YES/NO. Scores range from 0 to 100 points, with 0 indicating that the subject does not suffer from any health problems and 100 indicating that he or she suffers from all of them.
Independent values | All were measured at the start of the intervention and at week 24.
  Age and sex
Independent Values: Weight | The start of the intervention, week 6, week 9 and at week 24.
  Weight (Kilograms)
Independent Values: Height | The start of the intervention and at week 24.
  Height (Metre)
Independent Values: body mass index (BMI) | The start of the intervention, week 6, week 9 and at week 24.
  body mass index (BMI) (kg/m2).
Independent Values: general analytical and biochemical parameters | The start of the intervention and at 24/48 hours after surgery
  number of white blood cells and red blood cells, number of platelets, blood hemoglobin and hematocrit value in femtoliters.

CONTACTS AND LOCATIONS:
Overall Officials: IRENE MARIA IMLP LOPERA PAREJA, PRINCIPAL INVESTIGATOR, Principal Investigator — University of Jaen; IRENE MARIA IM LOPERA, Investigator, Principal Investigator — University of Jaen
Locations (1):
- Hospital Universitario Costa Del Sol, Marbella, Spain

IPD SHARING:
Plan to Share IPD: Yes
Plan for Sharing IPD from a Clinical Trial:
  1. Objective: Promote transparency, reproducibility, and new knowledge generation while safeguarding participant confidentiality.
  2. Ethical and legal aspects: Verify informed consent, de-identify data, and comply with regulations (e.g., GDPR, HIPAA).
  3. Preparation: Review and anonymize data, accompanied by key documentation (data dictionary, protocol, CSR).
  4. Infrastructure: Use secure platforms (e.g., Vivli, ClinicalStudyDataRequest) with access controls and traceability.
  5. Access: Review requests based on clear criteria; require data use agreements (DUA) and ethical commitment from researchers.
  6. Timeline: Share data 6-12 months after publication, available for 5-10 years.
  7. Oversight: Monitor requests and compliance; assess impact and adjust the plan based on feedback.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2025- January 2026
Access Criteria: Access Criteria for IPD Sharing:
  Research Purpose: Access is granted solely for valid scientific research that aligns with the objectives of the original study or advances medical knowledge.
  Application Requirements: Applicants must submit a detailed research proposal, including objectives, methodology, and justification for using the requested data.
  Researcher Qualifications: Access is limited to qualified researchers affiliated with recognized institutions.
  Data Use Agreement (DUA): Applicants must sign a DUA, agreeing to use the data only for the approved purpose, maintain confidentiality, and avoid re-identification of participants.
  Ethical Compliance: The research must have ethics committee approval and comply with relevant legal and regulatory standards.
  Transparency: Researchers must commit to publishing results in peer-reviewed journals or other scientific forums.

REFERENCES:
- [Background] Granicher P, Mulder L, Lenssen T, Fucentese SF, Swanenburg J, De Bie R, Scherr J. Exercise- and education-based prehabilitation before total knee arthroplasty: a pilot study. J Rehabil Med. 2024 Jan 8;56:jrm18326. doi: 10.2340/jrm.v56.18326. PMID 38192160
- [Background] Franz A, Ji S, Bittersohl B, Zilkens C, Behringer M. Impact of a Six-Week Prehabilitation With Blood-Flow Restriction Training on Pre- and Postoperative Skeletal Muscle Mass and Strength in Patients Receiving Primary Total Knee Arthroplasty. Front Physiol. 2022 Jun 14;13:881484. doi: 10.3389/fphys.2022.881484. eCollection 2022. PMID 35774280
- [Background] Swank AM, Kachelman JB, Bibeau W, Quesada PM, Nyland J, Malkani A, Topp RV. Prehabilitation before total knee arthroplasty increases strength and function in older adults with severe osteoarthritis. J Strength Cond Res. 2011 Feb;25(2):318-25. doi: 10.1519/JSC.0b013e318202e431. PMID 21217530
- [Background] McKay C, Prapavessis H, Doherty T. The effect of a prehabilitation exercise program on quadriceps strength for patients undergoing total knee arthroplasty: a randomized controlled pilot study. PM R. 2012 Sep;4(9):647-56. doi: 10.1016/j.pmrj.2012.04.012. Epub 2012 Jun 13. PMID 22698852
- [Background] Vitaloni M, Botto-van Bemden A, Sciortino Contreras RM, Scotton D, Bibas M, Quintero M, Monfort J, Carne X, de Abajo F, Oswald E, Cabot MR, Matucci M, du Souich P, Moller I, Eakin G, Verges J. Global management of patients with knee osteoarthritis begins with quality of life assessment: a systematic review. BMC Musculoskelet Disord. 2019 Oct 27;20(1):493. doi: 10.1186/s12891-019-2895-3. PMID 31656197
- [Background] Nguyen C, Boutron I, Roren A, Anract P, Beaudreuil J, Biau D, Boisgard S, Daste C, Durand-Zaleski I, Eschalier B, Gil C, Lefevre-Colau MM, Nizard R, Perrodeau E, Rabetrano H, Richette P, Sanchez K, Zalc J, Coudeyre E, Rannou F. Effect of Prehabilitation Before Total Knee Replacement for Knee Osteoarthritis on Functional Outcomes: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e221462. doi: 10.1001/jamanetworkopen.2022.1462. PMID 35262716
- [Background] Dong Y, Yan Y, Zhou J, Zhou Q, Wei H. Evidence on risk factors for knee osteoarthritis in middle-older aged: a systematic review and meta analysis. J Orthop Surg Res. 2023 Aug 29;18(1):634. doi: 10.1186/s13018-023-04089-6. PMID 37641050
- [Background] Jahic D, Omerovic D, Tanovic AT, Dzankovic F, Campara MT. The Effect of Prehabilitation on Postoperative Outcome in Patients Following Primary Total Knee Arthroplasty. Med Arch. 2018 Dec;72(6):439-443. doi: 10.5455/medarh.2018.72.439-443. PMID 30814777
- [Background] das Nair R, Mhizha-Murira JR, Anderson P, Carpenter H, Clarke S, Groves S, Leighton P, Scammell BE, Topcu G, Walsh DA, Lincoln NB. Home-based pre-surgical psychological intervention for knee osteoarthritis (HAPPiKNEES): a feasibility randomized controlled trial. Clin Rehabil. 2018 Jun;32(6):777-789. doi: 10.1177/0269215518755426. Epub 2018 Feb 9. PMID 29424236
- [Background] Chao J, Jing Z, Xuehua B, Peilei Y, Qi G. Effect of Systematic Exercise Rehabilitation on Patients With Knee Osteoarthritis: A Randomized Controlled Trial. Cartilage. 2021 Dec;13(1_suppl):1734S-1740S. doi: 10.1177/1947603520903443. Epub 2020 Feb 10. PMID 32037857
- [Background] Bennell KL, Nelligan RK, Kimp AJ, Schwartz S, Kasza J, Wrigley TV, Metcalf B, Hodges PW, Hinman RS. What type of exercise is most effective for people with knee osteoarthritis and co-morbid obesity?: The TARGET randomized controlled trial. Osteoarthritis Cartilage. 2020 Jun;28(6):755-765. doi: 10.1016/j.joca.2020.02.838. Epub 2020 Mar 19. PMID 32200051
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Koffel E, Kats AM, Kroenke K, Bair MJ, Gravely A, DeRonne B, Donaldson MT, Goldsmith ES, Noorbaloochi S, Krebs EE. Sleep Disturbance Predicts Less Improvement in Pain Outcomes: Secondary Analysis of the SPACE Randomized Clinical Trial. Pain Med. 2020 Jun 1;21(6):1162-1167. doi: 10.1093/pm/pnz221. PMID 31529104
- [Background] Alghadir AH, Anwer S, Sarkar B, Paul AK, Anwar D. Effect of 6-week retro or forward walking program on pain, functional disability, quadriceps muscle strength, and performance in individuals with knee osteoarthritis: a randomized controlled trial (retro-walking trial). BMC Musculoskelet Disord. 2019 Apr 9;20(1):159. doi: 10.1186/s12891-019-2537-9. PMID 30967128
- [Background] Gao B, Li L, Shen P, Zhou Z, Xu P, Sun W, Zhang C, Song Q. Effects of proprioceptive neuromuscular facilitation stretching in relieving pain and balancing knee loading during stepping over obstacles among older adults with knee osteoarthritis: A randomized controlled trial. PLoS One. 2023 Feb 13;18(2):e0280941. doi: 10.1371/journal.pone.0280941. eCollection 2023. PMID 36780435
- [Background] Ughi N, Prevete I, Ramonda R, Cavagna L, Filippou G, Manara M, Bortoluzzi A, Parisi S, Ariani A, Scire CA. The Italian Society of Rheumatology clinical practice guidelines for the diagnosis and management of gout. Reumatismo. 2019 Sep 23;71(S1):50-79. doi: 10.4081/reumatismo.2019.1176. PMID 31948193

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT06721897/Prot_SAP_ICF_000.pdf